CLINICAL TRIAL: NCT01586689
Title: Evaluating Alternative Aftercare Models for Ex-offenders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Professor, DePaul University, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OHEO1
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2014-09

CONDITIONS: Drug/Substance Abuse/Addiction; Alcohol Abuse/Addiction
Keywords: Oxford House; recovery; substance abuse; alcohol abuse; addiction
MeSH Terms: conditions — Behavior, Addictive; Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Safe Haven (Experimental): participants assigned to the Safe haven condition and agree to move into the A Safe Haven residential treatment facility
  Interventions: Behavioral: Safe Haven
- Usual aftercare (Experimental): participants assigned to the control condition, and may or may not seek treatment on their own
  Interventions: Behavioral: Usual aftercare
- Oxford House (Experimental): participants who were assigned to the Oxford House condition and agree to move into an Oxford House
  Interventions: Behavioral: Oxford House

INTERVENTIONS:
Behavioral: Oxford House — community-based recovery home for participants recovering from substance dependency
  Arms: Oxford House
Behavioral: Safe Haven — professionally-staffed treatment facility
  Arms: Safe Haven
Behavioral: Usual aftercare — control group - participants may or may not seek treatment on their own
  Arms: Usual aftercare

SUMMARY:
This study is examining the relative effects of alternative aftercare models for ex-offenders who are recovering from substance abuse/addiction. The study is a longitudinal, randomized field trial that assigns participants to one of three conditions: Oxford House, a professionally-run residential treatment facility, or a control condition that involves usual aftercare chosen by participants (which may include no treatment at all). Oxford Houses are self-run residential recovery homes based on the premise of mutual support. These homes do not involve professional treatment staff and the expenses (e.g. rent, utilities) are paid for by the residents. The hypothesis of this study is that Oxford House participants will have as good or better outcomes in terms of substance recovery, recidivism, and health in comparison to the participants who were assigned to the residential treatment facility, and better outcomes in comparison to the control group. In addition, the cost to government/tax payers will be substantially lower given that participants pay their own way.

ELIGIBILITY:
Inclusion Criteria:

* released from prison/jail in last 24 months
* recovering from alcohol or drug dependence

Exclusion Criteria:

* convicted of violent crime such as murder, aggravated assault
* currently using alcohol or drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2006-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Relapse/recovery - drug test and self report of alcohol use | last data collection point (wave 5, 2 years after recruitment)
  An assessment of each participant's drug/alcohol use as determined by a urine test and report of alcohol use
recidivism | last data collection point (wave 5, 2 years after recruitment)
  whether or not the participant has been re-incarcerated, as indicated by Illinois Department of Corrections data base
health | last data collection point (wave 5, 2 years after recruitment)
  participant health, such as hospitalization and other indicators as measured by the Addiction Severity Index (ASI) - Light. also measures substance use, employment, legal system involvement, family and social life, psychiatric status.

SECONDARY OUTCOMES:
Drug Taking Confidence Questionnaire (DTCQ) | every 6 months for 2 years
  confidence to avoid using drugs and alcohol in various situations;
Risk Behavior Survey | every 6 months for 2 years
  recent substance use and sexual behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Jason, PhD, Principal Investigator — DePaul University
Locations (1):
- DePaul University, Chicago, Illinois, United States

REFERENCES:
- [Background] Jason, L.A., Olson, B.D., Mueller, D.G., Walt, L., & Aase, D.M. (2010). Residential recovery homes/Oxford Houses In B. White & J. Kelly (eds.) Addiction Recovery Management: Theory, Research and Practice. (pp. 143-161). New York: Humana Press.
- [Background] Jason LA, Ferrari JR. Oxford House Recovery Homes: Characteristics and Effectiveness. Psychol Serv. 2010 May;7(2):92-102. doi: 10.1037/a0017932. PMID 20577571
- See also: DePaul Oxford House research project home page — http://condor.depaul.edu/ljason/oxford/